CLINICAL TRIAL: NCT02110901
Title: Multicenter, Double-Blind, Placebo-Controlled Study of PRT-201 Administered Immediately After Radiocephalic Arteriovenous Fistula Creation in Patients With Chronic Kidney Disease
Brief Title: A Study of PRT-201 Administered Immediately After Radiocephalic Arteriovenous Fistula(AVF) Creation in Patients With Chronic Kidney Disease (CKD) (PATENCY-1)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Proteon Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PRT-201-310
Record Dates: First submitted 2014-04-02; First posted 2014-04-10 (Estimated); Results first posted 2019-07-09 (Actual); Last update posted 2019-07-09 (Actual); Status verified 2019-06

CONDITIONS: Chronic Kidney Disease
Keywords: radiocephalic; arteriovenous fistula; AVF; hemodialysis; PRT-201; vascular access; kidney; renal; vonapanitase; PATENCY-1
MeSH Terms: conditions — Renal Insufficiency, Chronic; Arteriovenous Fistula | interventions — cholesterol-binding protein

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- PRT-201 (Active Comparator): PRT-201 administered at the time of radiocephalic fistula creation
  Interventions: Drug: PRT-201
- Placebo (Placebo Comparator): Placebo administered at the time of radiocephalic fistula creation. The placebo is identical in appearance and composition to PRT-201 but lacks the active ingredient.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: PRT-201
  Other Names: vonapanitase
  Arms: PRT-201
Drug: Placebo
  Arms: Placebo

SUMMARY:
This research study is designed to assess the safety and effectiveness of an experimental drug called PRT-201 in patients both receiving or expecting to receive dialysis who have chronic kidney disease and who are undergoing surgery to create a new access point to their bloodstream for hemodialysis. PRT-201 is a protein that has been shown in previous research studies to help keep vessels patent when applied to the outside surface of the blood vessels (arteries and veins) in patients who undergo surgery to create an arteriovenous fistula (AVF). The purpose of this study is to determine whether PRT-201 when applied to a limited segment of your blood vessel (about 2 inches) immediately after surgery is safe and improves the patency of your AVF.

ELIGIBILITY:
Inclusion Criteria:

1. Age of at least 18 years.
2. Life expectancy of at least 6 months.
3. Diagnosis of Chronic Kidney Disease (CKD).
4. Planned creation of a new radiocephalic arteriovenous fistula (AVF)-revision of an existing AVF is not eligible.
5. Ability to understand and comply with the requirements of the entire study and to communicate with the study team.
6. Written informed consent using a document that has been approved by the Institutional Review Board (IRB).
7. If female and of childbearing potential (premenopausal and not surgically sterile) must have a negative serum pregnancy test at the screening visit (Visit 1) and be willing to use contraception from the time of the screening visit to 2 weeks following study drug administration. Acceptable methods of birth control include abstinence, barrier methods, hormones, or intra uterine device.

Exclusion Criteria:

1. Malignancy or treatment for malignancy within the previous 12 months with the exception of the following cancers if they have been resected: localized basal cell or squamous cell skin cancer, or any cancer in situ.
2. Presence of any significant medical condition that might significantly confound the collection of safety and efficacy data in this study.
3. Previous treatment with PRT 201.
4. Treatment with any investigational drug within the previous 30 days or investigational antibody therapy within the previous 90 days prior to signing informed consent.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 349 (Actual)
Dates: Start 2014-07 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2018-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (35):
- United States (35):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - AKDHC Medical Research Services , LLC, Phoenix, Arizona
  - AKDHC Medical Research Services, LLc, Tucson, Arizona
  - Alliance Research Center, Laguna Hills, California
  - VA Medical Center Long Beach, Long Beach, California
  - Keck University Hospital at USC, Los Angeles, California
  - Kaiser Permanente Medical Center, San Diego, California
  - California Institute of Renal Research, San Diego, California
  - UCSF Division of Vascular & Endovascular Surgery, San Francisco, California
  - Rush Medical Center, Chicago, Illinois
  - Renal Care Associates, Peoria, Illinois
  - Lutheran Hospital Network of Indiana, Fort Wayne, Indiana
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - University of Louisville, Louisville, Kentucky
  - Tulane University, New Orleans, Louisiana
  - Louisiana State University Health Sciences Center, Shreveport, Louisiana
  - Maine Medical Center, Portland, Maine
  - University of Maryland, Baltimore, Maryland
  - University of Maryland Shore Medical Center at Easton, Easton, Maryland
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts
  - University of Massachusetts Medical Center, Worcester, Massachusetts
  - Mount Sinai Medical Center, New York, New York
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Duke University, Durham, North Carolina
  - W.G. Hefner VA Medical Center, Salisbury, North Carolina
  - Wake Forest, Winston-Salem, North Carolina
  - University of Cincinnati Medical Center, Cincinnati, Ohio
  - University of Cincinnati, Cincinnati, Ohio
  - Ohio State University, Columbus, Ohio
  - The University of Oklahoma College of Medicine, Tulsa, Oklahoma
  - Lehigh Valley Health Network, Allentown, Pennsylvania
  - VA Pittsburg Healthcare System, Pittsburgh, Pennsylvania
  - The Methodist Hospital, Houston, Texas
  - Lake Washington Vascular Center, Bellevue, Washington

REFERENCES:
- [Derived] Heindel P, Fitzgibbon JJ, Secemsky EA, Belkin M, Ozaki CK, Hussain MA. Evaluating the effectiveness of systemic heparin during arteriovenous fistula creation by emulating a target trial. Am J Epidemiol. 2025 Mar 4;194(3):651-658. doi: 10.1093/aje/kwae098. PMID 38825327
- [Derived] Heindel P, Fitzgibbon JJ, Feliz JD, Hentschel DM, Burke SK, Al-Omran M, Bhatt DL, Belkin M, Ozaki CK, Hussain MA. Evaluating national guideline concordance of recurrent interventions after radiocephalic arteriovenous fistula creation. J Vasc Surg. 2023 Apr;77(4):1206-1215.e2. doi: 10.1016/j.jvs.2022.12.017. Epub 2022 Dec 22. PMID 36567000
- [Derived] Bleyer AJ, Scavo VA, Wilson SE, Browne BJ, Ferris BL, Ozaki CK, Lee T, Peden EK, Dixon BS, Mishler R, O'Connor TP, Kidd K, Burke SK; PATENCY-1 Investigators. A randomized trial of vonapanitase (PATENCY-1) to promote radiocephalic fistula patency and use for hemodialysis. J Vasc Surg. 2019 Feb;69(2):507-515. doi: 10.1016/j.jvs.2018.04.068. PMID 30683197

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 349 patients signed informed consent; 313 patients were randomized; 311 were treated
Pre-assignment Details: Participants were excluded from participation if they did not have a radiocephalic AVF created at the time of surgery.
Groups:
- Vonapanitase: Vonapanitase administered at the time of radiocephalic fistula creation
- Placebo: Placebo administered at the time of radiocephalic fistula creation
Period: Overall Study
Arm/Group | Vonapanitase | Placebo
Started | 209 | 102
Completed | 179 | 88
Not Completed | 30 | 14
Not completed — Death | 6 | 3
Not completed — Lost to Follow-up | 12 | 8
Not completed — Withdrawal by Subject | 7 | 3
Not completed — received a kidney transplant | 5 | 0

BASELINE CHARACTERISTICS:
Groups:
- Vonapanitase; Placebo: Single application administered over 10 minutes at the time of fistula creation.
- Total: Total of all reporting groups
Arm/Group | Vonapanitase | Placebo | Total
Number analyzed (Participants) | 209 | 102 | 311
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 143 | 71 | 214
  >=65 years | 66 | 31 | 97
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 36 | 26 | 62
  Male | 173 | 76 | 249
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 29 | 19 | 48
  Not Hispanic or Latino | 180 | 83 | 263
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 0 | 2
  Asian | 6 | 5 | 11
  Native Hawaiian or Other Pacific Islander | 2 | 0 | 2
  Black or African American | 55 | 19 | 74
  White | 138 | 71 | 209
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 6 | 7 | 13
Region of Enrollment [Number; unit: participants]
  United States | 209 | 102 | 311

OUTCOME MEASURES:

1. Primary Outcome: Time to AVF Primary Unassisted Patency
Description: Primary unassisted patency defined as the time from AVF creation until the first occurrence of either access thrombosis or procedure to restore or maintain patency.
Time Frame: Days from AVF creation until the first occurrence of either access thrombosis or procedure to restore or maintain patency, assessed up to 1 year
Population: Full analysis set includes any patient who was randomized.
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Vonapanitase | Placebo
Number analyzed (Participants) | 210 | 103
Days | 214 [163 to 322] | 171 [126 to 285]
Statistical Analysis 1: Comparison: Vonapanitase vs Placebo; Test type: Superiority; p = 0.254, Log Rank; Hazard Ratio (HR) = 0.83, 95% CI 2-sided [0.61 to 1.14]

2. Primary Outcome: Kaplan-Meier Estimate of Secondary AVF Patency
Description: Kaplan-Meier Estimate of median time from AVF creation until AVF abandonment (secondary patency)
Time Frame: Median time from AVF creation until AVF abandonment (secondary patency), assessed up to 1 year
Population: Full analysis set included all patients who were randomized
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Vonapanitase | Placebo
Number analyzed (Participants) | 210 | 103
days | NA [NA to NA] — The median time to AVF abandonment based on Kaplan-Meier estimates was not reached in this trial | NA [NA to NA] — The median time to AVF abandonment based on Kaplan-Meier estimates was not reached in this trial
Statistical Analysis 1: Comparison: Vonapanitase vs Placebo; Test type: Superiority; p = 0.048, Log Rank; Hazard Ratio (HR) = 0.66, 95% CI 2-sided [0.43 to 1.00]

3. Other Pre Specified Outcome: Number of Participants With Unassisted AVF Maturation by Ultrasound
Description: AVF maturation is defined as average cephalic vein lumen diameter >= 4 mm and an outflow vein volume blood flow >= 500 mL/min by ultrasound without prior primary unassisted patency loss.
Time Frame: Assessed 3 months after AVF creation
Population: Full analysis set includes any patient who was randomized
Measure: Count of Participants; unit: Participants
Arm/Group | Vonapanitase | Placebo
Number analyzed (Participants) | 210 | 103
Participants
  With Unassisted AVF Maturation | 132 | 55
  Without Unassisted AVF Maturation | 78 | 48
Statistical Analysis 1: Comparison: Vonapanitase vs Placebo; Test type: Superiority; p = 0.109, Chi-squared

4. Other Pre Specified Outcome: Number of Participants With Unassisted AVF Use for Hemodialysis
Description: Unassisted AVF use for hemodialysis is defined as continuous use of the AVF for hemodialysis without prior primary unassisted patency loss. Use of the AVF for hemodialysis is defined as the ability of the study AVF to be successfully cannulated and used for hemodialysis for a minimum of 90 days or at least 30 days prior to a patient's last visit, if hemodialysis was not initiated at least 90 days prior to the last visit. Non-use of the AVF for hemodialysis is defined as an abandoned fistula prior to use; or if hemodialysis is recorded on 2 consecutive visits and there is no cannulation date or duration of use is less than 90 days. The patients who are not categorized as having use or non-use of the AVF by the rules described above have insufficient data to determine use for hemodialysis and will be categorized as having indeterminate use.
Time Frame: Assessed at 12 months
Population: Patients with unassisted use or non-use of their AVF for hemodialysis. Patients with indeterminate use of their AVF were excluded.
Measure: Count of Participants; unit: Participants
Arm/Group | Vonapanitase | Placebo
Number analyzed (Participants) | 158 | 72
Participants
  New AVF Used Unassisted | 62 | 18
  New AVF Not Used or Assisted Use | 96 | 54
Statistical Analysis 1: Comparison: Vonapanitase vs Placebo; Test type: Superiority; p = 0.035, Chi-squared

ADVERSE EVENTS:
Time Frame: All adverse events through Week 6 were collected. Week 6-Month 12 only AEs associated with the AVF extremity were collected.
Groups:
- Vonapanitase: Vonapanitase administered at the time of radiocephalic fistula creation
  Vonapanitase
- Placebo: Placebo administered at the time of radiocephalic fistula creation. The placebo is identical in appearance and composition to PRT-201 but lacks the active ingredient.
  Placebo
Arm/Group | Vonapanitase | Placebo
All-Cause Mortality (participants affected / at risk) | 7/209 | 4/102
Serious Adverse Events (participants affected / at risk) | 29/209 | 15/102
Other Adverse Events (participants affected / at risk) | 149/209 | 84/102
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Vonapanitase (N=209) | Placebo (N=102)
Coagulopathy (Blood and lymphatic system disorders) | 0 | 1
Cardiac Arrest (Cardiac disorders) | 1 | 1
Cardiac Failure Congestive (Cardiac disorders) | 1 | 0
Coronary Artery Disease (Cardiac disorders) | 1 | 0
Pulseless Electrical Activity (Cardiac disorders) | 1 | 0
Supraventricular Tachycardia (Cardiac disorders) | 1 | 0
Myocardial Infarction (Cardiac disorders) | 0 | 1
Acute Myocardial Infarction (Cardiac disorders) | 0 | 1
Colitis (Gastrointestinal disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0
Death (General disorders) | 1 | 0
Chest Pain (General disorders) | 0 | 1
Systemic Inflammatory Response Syndrome (General disorders) | 0 | 1
Sepsis (Infections and infestations) | 2 | 0
Arthritis Bacterial (Infections and infestations) | 1 | 0
Cellulitis (Infections and infestations) | 1 | 0
infection (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 0 | 3
Anaemia (Blood and lymphatic system disorders) | 1 | 0
Arteriovenous Fistula Thrombosis (Injury, poisoning and procedural complications) | 2 | 1
Injury (Injury, poisoning and procedural complications) | 1 | 0
Limb Injury (Injury, poisoning and procedural complications) | 1 | 0
Fluid Overload (Metabolism and nutrition disorders) | 2 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 2 | 0
Gout (Metabolism and nutrition disorders) | 0 | 1
Ketoacidosis (Metabolism and nutrition disorders) | 0 | 1
Hypoxic-Ischaemic Encephalopathy (Nervous system disorders) | 1 | 0
Metabolic Encephalopathy (Nervous system disorders) | 1 | 1
Major Depression (Psychiatric disorders) | 1 | 0
Renal Failure Acute (Renal and urinary disorders) | 1 | 0
Renal Failure Chronic (Renal and urinary disorders) | 0 | 1
Chronic Obstructive Pulmonary Disease (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Acute Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Haemoptyis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Diabetic Foot (Skin and subcutaneous tissue disorders) | 1 | 0
Decubitus Ulcer (Skin and subcutaneous tissue disorders) | 0 | 1
Deep Vein Thrombosis (Vascular disorders) | 1 | 0
Hypertensive Crisis (Vascular disorders) | 1 | 1
Shock (Vascular disorders) | 1 | 0
Steal Syndrome (Vascular disorders) | 1 | 0
Vascular Stenosis (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Vonapanitase (N=209) | Placebo (N=102)
Procedural Pain (Injury, poisoning and procedural complications) | 10 | 6
Arteriovenous fistula thrombosis (Injury, poisoning and procedural complications) | 41 | 27
Hypoaesthesia (Nervous system disorders) | 11 | 5
Vascular Stenosis (Vascular disorders) | 80 | 41
Haematoma (Vascular disorders) | 7 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No